CLINICAL TRIAL: NCT05225194
Title: Prospective Study for the Assessment of Long-term Impact of COVID-19 Among COVID-19 Patients With Acute Respiratory Distress Syndrome in Brazil
Brief Title: Long-term Impact of COVID-19 Among COVID-19 Patients With Acute Respiratory Distress Syndrome in Brazil
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Other Study IDs: Pos-COVID Brasil 3
Record Dates: First submitted 2022-02-01; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; ARDS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 ARDS survivors: Survivors of hospitalization due to ARDS caused by SAS-CoV-2.
  Interventions: Other: COVID-19; Other: ARDS
- Non-COVID-19 ARDS survivors: Survivors of hospitalization due to ARDS caused by other etiologies than SARS-CoV-2.
  Interventions: Other: ARDS
- Family controls: Family controls of participants with ARDS (either due to COVID-19 or other etiologies) without history of COVID-19 or hospitalization in the last 12 months.

INTERVENTIONS:
Other: COVID-19 — SARS-CoV-2 infection
  Groups: COVID-19 ARDS survivors
Other: ARDS — Acute respiratory distress syndrome
  Groups: COVID-19 ARDS survivors; Non-COVID-19 ARDS survivors

SUMMARY:
The present multicenter prospective observational study aims to assess the long-term effects of COVID-19 on patients with Acute Respiratory Distress Syndrome (ARDS).

This is a hybrid design study with components of cohort and case-control designs. Survivors of hospitalization due to ARDS caused by SARS-CoV-2, survivors of hospitalization due to ARDS caused by other etiologies not associated with SARS-CoV-2, and family controls without history of COVID-19 or hospitalization will be followed up for a period of 6 months.

ELIGIBILITY:
COHORT OF SURVIVORS OF ARDS CAUSED BY COVID-19

Inclusion Criteria:

* Age ≥18 years;
* Hospitalization due to COVID-19;
* Positive polymerase chain reaction (PCR) test for SARS-CoV-2;
* Diagnosis of ARDS during hospitalization according to the Berlin definition;
* Expected to survive and be discharged directly home from the hospital.

Exclusion Criteria:

* Severe comorbidity with life expectancy less than 3 months;
* Unavailability to attend the study follow-up appointment;
* Death during hospitalization;
* Absence of proxy for patients with communication difficulties;
* Refusal or withdrawal of agreement to participate.

COHORT OF SURVIVORS OF ARDS CAUSED BY OTHER ETIOLOGIES NOT ASSOCIATED WITH COVID-19

Inclusion Criteria:

* Age ≥18 years;
* Hospitalization;
* Diagnosis of ARDS during hospitalization according to the Berlin definition;
* Expected to survive and be discharged directly home from the hospital.

Exclusion Criteria:

* Severe comorbidity with life expectancy less than 3 months;
* Unavailability to attend the study follow-up appointment;
* Death during hospitalization;
* History of SARS-CoV-2 infection within the last 12 months;
* Absence of proxy for patients with communication difficulties;
* Refusal or withdrawal of agreement to participate.

FAMILY CONTROLS

Inclusion Criteria:

* Age ≥18 years;
* Family member of a enrolled participant (either from the COVID-19 ARDS cohort or from the non-COVID-19 ARDS cohort)

Exclusion Criteria:

* Severe comorbidity with life expectancy less than 3 months;
* Unavailability to attend the study follow-up appointment;
* History of SARS-CoV-2 infection within the last 12 months;
* History of non-elective hospitalization due to medical condition within the last 12 months;
* Refusal or withdrawal of agreement to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Survivors of hospitalization due to ARDS caused by SARS-CoV-2, survivors of hospitalization due to ARDS caused by other etiologies not associated with SARS-CoV-2, and family controls without history of COVID-19 or hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Diffusion capacity for carbon monoxide | The outcome will be assessed 6 months after enrollment
  Proportion of participants with diffusion capacity for carbon monoxide < 80% of predicted

SECONDARY OUTCOMES:
Physical functional status | The outcome will be assessed at 3 and 6 months after enrollment
  Physical functional status as assessed by the modified Barthel index (score ranges from 0 to 100; higher scores indicate less functional dependence)
Instrumental Activities of Daily Living | The outcome will be assessed at 3 and 6 months after enrollment
  The outcome will be assessed using the Lawton & Brody Instrumental Activities of Daily Living Scale (the score ranges from 0 to 8, with higher scores indicating less dependence)
Muscular function and strength | The outcome will be assessed at 3 and 6 months after enrollment
  Muscular function and strength as assessed by Strength, assistance with walking, rising from a chair, climbing stairs, and falls (SARC-F) questionnaire. Scale scores range from 0 (best) to 10 (worst)
Score of dyspnea | The outcome will be assessed at 3 and 6 months after enrollment
  The outcome will be assessed using the modified medical research council dyspnea scale. Scores ranges from 0 to 4, with higher scores indicating worse symptoms.
Utility score of health related quality of life | The outcome will be assessed at 3 and 6 months after enrollment
  The outcome will be assessed using the Brazilian version of the Euroqol-5D-3L (EQ-5D3L) questionnaire. The utility score derived from the EQ5D-3L ranges from 0 (death) to 1 (perfect health).
Radiologic patterns of intersticial lung disease | The outcome will be assessed at 6 months after enrollment
  Radiologic patterns of intersticial lung disease as assessed by high resolution computed tomography chest scan.
Radiologic patterns of myocarditis sequalae | The outcome will be assessed at 6 months after enrollment
  Radiologic patterns of myocarditis sequalae as assessed by cardiac magnetic resonance imaging
Radiologic patterns of sarcopenia | The outcome will be assessed at 6 months after enrollment
  Radiologic patterns of sarcopenia as assessed by high resolution computed tomography chest scan.
Incidence of major cardiovascular events | The outcome will be assessed at 3 and 6 months after enrollment
  Incidence of major cardiovascular events (composite endpoint of non-fatal stroke, non-fatal acute myocardial infarction, or cardiovascular death)
Incidence of thromboembolic events | The outcome will be assessed at 3 and 6 months after enrollment
  Incidence of thromboembolic events (composite endpoint of pulmonary embolism and deep venous thrombosis)
Incidence of all-cause mortality | The outcome will be assessed at 3 and 6 months after enrollment
  Incidence of all-cause mortality
Percentage of predicted peak oxygen consumption | The outcome will be assessed at 6 months after enrollment
  Percentage of predicted peak oxygen consumption as assessed by treadmill cardiopulmonary exercise cardiopulmonary exercise
Peak oxygen consumption | The outcome will be assessed at 6 months after enrollment
  Peak oxygen as assessed by treadmill cardiopulmonary exercise
Peak oxygen pulse | The outcome will be assessed at 6 months after enrollment
  Peak oxygen pulse as assessed by treadmill cardiopulmonary exercise
Oxygen uptake efficiency slope | The outcome will be assessed at 6 months after enrollment
  Oxygen uptake efficiency slope as assessed by treadmill cardiopulmonary exercise
Minute ventilation/carbon dioxide production slope ratio | The outcome will be assessed at 6 months after enrollment
  Minute ventilation/carbon dioxide production slope as assessed by treadmill cardiopulmonary exercise
Forced vital capacity | The outcome will be assessed at 6 months after enrollment
  Forced expiratory capacity as assessed by spirometry
Forced expiratory volume in one second | The outcome will be assessed at 6 months after enrollment
  Forced expiratory volume in one second as assessed by spirometry
Forced expiratory volume in one second/ Forced vital capacity ratio | The outcome will be assessed at 6 months after enrollment
  Forced expiratory volume in one second/ Forced vital capacity ratio as assessed by spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Regis G Rosa, MD, PhD, Principal Investigator — Hospital Moinhos de Vento